CLINICAL TRIAL: NCT03941301
Title: Light Therapy on Major Depression Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mackay Memorial Hospital (Other)
Collaborators: National Tsing Hua University,Taiwan (Other); Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 18MMHIS114e
Record Dates: First submitted 2019-03-27; First posted 2019-05-07 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Depressive Disorder
MeSH Terms: conditions — Depressive Disorder | interventions — Phototherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bright treatment light (Experimental)
  Interventions: Device: Light therapy
- Red light (Placebo Comparator)
  Interventions: Device: Light therapy

INTERVENTIONS:
Device: Light therapy — Participants will be exposed to bright treatment light or red light 30 minutes every day for 4 weeks.

SUMMARY:
Background:

Major depression disorder is a common psychological disease. It is the second-ranked cause of disability worldwide. The pathophysiology is not yet understood. The main theory is monoaminergic theory based on the effect of monoaminergic drugs. Current treatment includes psychotherapy, medication and electroconvulsive therapy. The onset of action for antidepressant is often slow, therefore strategies to improve the outcome are important. Bright light therapy has been found to be effective in reducing the severity of depression not only in seasonal affective disorder but also in other affective disorder. Previous meta-analyses of light therapy for non-seasonal major depression, however, has yielded conflicting evidence for efficacy.

Purpose:

1. To investigate possible imaging biomarkers of major depression disorder
2. To evaluate the effect of light therapy on depression

Materials and Methods:

This prospective study will recruit 100 patients, randomized into 2 study groups: (1) antidepressant plus treatment light, and (2) antidepressant plus placebo light. All patients will accept a thorough psychological evaluation (including Hamilton Depression Rating Scale, Montgomery-Asberg Depression Rating Scale, Clinical Global Impression-Severity and Patient Health Questionnaire-9 items) at baseline and at the 1st, 2nd, 4th, 8th week during the 8-week experiment intervention, by a blind assessor. Morningness- Eveningness Questionnaire-Self-Assessment Version (MEQ-SA) was only evaluated at baseline. Adverse events were evaluated at baseline, 2nd,4th,8th weeks. MRI study will be arranged at baseline and in 4-week experiment.

Predicted Results and Influence:

1. To evaluate the additional effect of the treatment light on depression disorder
2. To compare the difference of functional magnetic resonance imaging(fMRI), structural MRI among the two groups and between the patients with and without treatment effect in order to detect imaging biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Fulfill diagnosis of Major depression disorder based on Diagnostic and Statistical Manual of Mental Disorders(DSM-V) for at least 6 weeks and under medication treatment for at least 4 weeks.
2. at least 20 years old
3. Hamilton Depression Rating Scale(HAMD-17) >= 13
4. No medication change for at least 4 weeks and no medication change will be considered in the next 8 weeks.
5. Agree to participate in this study and sign the permit.

Exclusion Criteria:

1. Seasonal depression disorder
2. Other psychological or neurological disorder
3. Drug or alcohol abuse within 30 days
4. Visual problem
5. Light-induced seizure or migraine
6. Contraindication for MRI study
7. Severe illness and might be admitted in the near future
8. Might have a long trip in the near future

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Hamilton Depression Rating Scale(HAM-D) at 1,2,4,8 weeks | 1,2,4,8 weeks.
  Determine severity of depression (scores: 0-50)
  1. Depressed Mood (sadness, hopeless, helpless, worthless) (0-4 scores)
  2. Feelings of Guilt(0-4 scores)
  3. Suicide(0-4 scores)
  4. Insomnia - Early(0-2 scores)
  5. Insomnia - Middle(0-2 scores)
  6. Insomnia - Late(0-2 scores)
  7. Work and Activities(0-4 scores)
  8. Retardation (slowness of thought and speech; impaired ability to concentrate; decreased motor activity)(0-4 scores)
  9. Agitation(0-2 scores)
  10. Anxiety - Psychic(0-4 scores)
  11. Anxiety - Somatic(0-4 scores)
  12. Somatic Symptoms - Gastrointestinal(0-2 scores)
  13. Somatic Symptoms - General(0-2 scores)
  14. Genital Symptoms(0-2 scores)
  15. Hypochondriasis(0-4 scores)
  16. Loss of Weight(0-2 scores)
  17. Insight(0-2 scores)
  Scores below 7 generally represent the absence or remission of depression. Scores between 7-17 represent mild depression. Scores between 18-24 represent moderate depression. Scores 25 and above represent severe depression.
Change from Baseline Montgomery-Asberg Depression Rating Scale(MADRS) at 1,2,4,8 weeks | 1,2,4,8 weeks.
  Higher MADRS score indicates more severe depression, and each item yields a score of 0 to 6. The overall score ranges from 0 to 60.
  The questionnaire includes questions on the following symptoms
  1. Apparent sadness 2. Reported sadness 3. Inner tension 4. Reduced sleep 5. Reduced appetite 6. Concentration difficulties 7. Lassitude 8. Inability to feel 9. Pessimistic thoughts 10. Suicidal thoughts
  0 to 6 - normal /symptom absent 7 to 19 - mild depression 20 to 34 - moderate depression >34 - severe depression
Change from Baseline Clinical Global Impression-Severity(CGI-S) at 1,2,4,8 weeks | 1,2,4,8 weeks.
  The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Possible ratings are:
  1. Normal, not at all ill
  2. Borderline mentally ill
  3. Mildly ill
  4. Moderately ill
  5. Markedly ill
  6. Severely ill
  7. Among the most extremely ill patients
Change from Baseline Patient Health Questionnaire(PHQ-9) at 1,2,4,8 weeks | 1,2,4,8 weeks.
  Depression screening by a nine-item in adults
  Over the last two weeks, how often have you been bothered by any of the following problems? (Scores: 0-27) 0:Not at all, 1:Several days, 2:More than half the days, 3:Nearly every day
  1. Little interest or pleasure in doing things
  2. Feeling down, depressed, or hopeless
  3. Trouble falling or staying asleep, or sleeping too much
  4. Feeling tired or having little energy
  5. Poor appetite or overeating
  6. Feeling bad about yourself, or that you are a failure, or have let yourself or your family down
  7. Trouble concentrating on things, such as reading the newspaper or watching television
  8. Moving or speaking so slowly that other people could have noticed? Or the opposite, being so fidgety or restless that you have been moving around a lot more than usual
  9. Thoughts that you would be better off dead or of hurting yourself in some way
  0-4:No depression, 5-9:Mild, 10-14:Moderate, 15-19:Moderately severe, 20-27: Severe

SECONDARY OUTCOMES:
functional MRI | 4 weeks
  Compare brain resting-state functional MRI change between these two arms.
  Including measures brain activity by detecting changes associated with blood flow and difference of Resting State Network which is a functionally connected neural network of apparent brain states.
  Increased strength of the activities or resting state network indicates neural activities are elevated within the regions of the brain or the network.
  Decreased strength of the activities or resting state network indicates neural activities are diminished within the regions of the brain or the network.
Diffusion Tensor Imaging of MRI | 4 weeks
  Compare brain Diffusion Tensor Imaging between these two arms.
  Evaluation the connection or fiber tracts between regions of the brain. Increased strength means enhanced connection between neuronal regions of the brain.
  Decreased strength means decreased connection between neuronal regions of the brain.

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Chao Huang, Principal Investigator — Mackay Memorial Hospital
Locations (1):
- Mackay Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang CC, Huang HC, Lin CJ, Hsu CC, Lee CS, Hsu YH, Chen TL, Liao WH, Wu YH, Yang FG, Liu SI. Subclinical alterations of resting state functional brain network for adjunctive bright light therapy in nonseasonal major depressive disorder: A double blind randomized controlled trial. Front Neurol. 2022 Nov 9;13:979500. doi: 10.3389/fneur.2022.979500. eCollection 2022. PMID 36438959